CLINICAL TRIAL: NCT01158521
Title: A Phase II Study of Pazopanib to Enable Partial Nephrectomy
Brief Title: Pazopanib Hydrochloride Before Surgery in Treating Patients With Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4809; NCI-2010-01392 (Other: NCI/CTRP)
Record Dates: First submitted 2010-07-01; First posted 2010-07-08 (Estimated); Results first posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Clear Cell Renal Cell Carcinoma; Stage I Renal Cell Cancer; Stage II Renal Cell Cancer; Stage III Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive oral pazopanib hydrochloride once daily for up to 18 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo either partial or radical nephrectomy at least 7 days after completion of pazopanib hydrochloride.
  Interventions: Drug: pazopanib hydrochloride; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Drug: pazopanib hydrochloride — Oral pazopanib hydrochloride once daily for up to 18 weeks in the absence of disease progression or unacceptable toxicity.
  Other Names: GW786034; Votrient
Procedure: therapeutic conventional surgery — Patients undergo either partial or radical nephrectomy at least 7 days after completion of pazopanib hydrochloride.

SUMMARY:
RATIONALE: Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving pazopanib hydrochloride before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well pazopanib hydrochloride works when given before surgery in treating patients with kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the rate of partial nephrectomy in patients with primary renal tumors otherwise requiring radical nephrectomy after neoadjuvant pazopanib treatment.

SECONDARY OBJECTIVES:

I. To determine the safety, tumor diameter/volume change, conversion of hilar to non-hilar tumors and surgical morbidity of neoadjuvant pazopanib for renal cell carcinoma (RCC).

OUTLINE:

Patients receive oral pazopanib hydrochloride once daily for up to 18 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo either partial or radical nephrectomy at least 7 days after completion of pazopanib hydrochloride.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion

* Histologically or cytologically proven renal carcinoma with a clear cell component
* Need for optimized partial nephrectomy based on one or more of the following criteria (all applicable criteria should be recorded and one criterion designated as the primary reason):

  * Functional or anatomic solitary kidney, bilateral tumors, or pre-existing chronic kidney disease (CKD; estimated glomerular filtration rate (GFR) by Cockcroft-Gault formula < 60 mL/min) and tumor amenable to partial nephrectomy, but partial nephrectomy would result in estimated GFR < 30 mL/min; this estimation will be based on current estimated GFR, nuclear renal scan to estimate relative renal function (if 2 kidneys), tumor location(s), and amount of normal renal parenchyma that would need to be removed with nephrectomy
  * Radical nephrectomy is required for tumor excision; however, it would result in estimated GFR < 30 mL/min; this estimation will be based on current estimated GFR, nuclear renal scan to estimate relative renal function (if 2 kidneys), tumor location(s), and amount of normal renal parenchyma that would need to be removed with radical nephrectomy
  * Greater than 30% likelihood that a partial nephrectomy would be associated with a high risk of significant morbidity (e.g. hemorrhage) due to proximity to the renal hilum (within 3 mm of main renal artery, renal vein or their primary branches) and/or other anatomic factors as determined by the operating surgeon
  * Renal nephrometry score of 10-12
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Karnofsky >= 70%
* Serum aspartate transaminase (AST; serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 x laboratory upper limit of normal (ULN)
* Serum alanine transaminase (ALT; serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x laboratory upper limit of normal (ULN)
* Total serum bilirubin =< 1.5 x ULN
* Absolute neutrophil count (ANC) >= 1500/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 9.0 g/dL (no transfusion permitted within 1 week)
* Serum creatinine =< 2.5 mg/dL
* Urine to protein to creatinine (UPC) ratio < 1; if UPC > 1, then a 24-hour urine protein must be assessed; subjects must have a 24-hour urine protein value < 1g to be eligible
* Prothrombin time (PT) or international normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.2 X upper limit of normal (ULN)
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures; subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow up
* A female is eligible to enter and participate in this study if she is of:
* Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had: a hysterectomy; a bilateral oophorectomy (ovariectomy); a bilateral tubal ligation; is post-menopausal
* Subjects not using hormone replacement therapy (HRT) must have experienced total cessation of menses for >= 1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone (FSH) value > 40 mIU/mL and an estradiol value < 40pg/mL (< 140 pmol/L)
* Subjects using HRT must have experienced total cessation of menses for >= 1 year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT
* Childbearing potential, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception; GlaxoSmithKlein (GSK) acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows: an intrauterine device with a documented failure rate of less than 1% per year; vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female; complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product; or double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide)

Exclusion

* Prior systemic treatment for RCC
* Evidence of any distant metastatic disease
* Evidence of bleeding diathesis or coagulopathy; patients with hematuria from the primary renal tumor are eligible provided all other eligibility criteria are met
* History of any one or more of the following cardiovascular conditions within the past 6 months: cardiac angioplasty or stenting; myocardial infarction; unstable angina; coronary artery bypass graft surgery; symptomatic peripheral vascular disease
* Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
* Prolongation of corrected QT interval (QTc) > 480 msecs
* Hypertension that cannot be controlled by medications to < 160/90 mmHg
* History of cerebrovascular accident, pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months (Note: subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible)
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major)
* Hemoptysis within 6 weeks of first dose of study drug
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures
* Unable or unwilling to discontinue use of prohibited medications for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study
* Clinically significant gastrointestinal abnormalities that may increase the risk for GI bleeding including, but not limited to: active peptic ulcer disease; known intraluminal metastatic lesion/s with suspected bleeding; inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation; history of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to: malabsorption syndrome; major resection of the stomach or small bowel
* Prior major surgery or trauma (NOT including biopsy of renal mass; also procedures such as catheter placement not considered to be major) within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer
* Presence of uncontrolled infection
* Other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the patient inappropriate for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Rini, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Lane BR, Derweesh IH, Kim HL, O'Malley R, Klink J, Ercole CE, Palazzi KL, Thomas AA, Rini BI, Campbell SC. Presurgical sunitinib reduces tumor size and may facilitate partial nephrectomy in patients with renal cell carcinoma. Urol Oncol. 2015 Mar;33(3):112.e15-21. doi: 10.1016/j.urolonc.2014.11.009. Epub 2014 Dec 19. PMID 25532471

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: Patients receive oral pazopanib hydrochloride once daily for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo either partial or radical nephrectomy at least 7 days after completion of pazopanib hydrochloride.
  pazopanib hydrochloride: Oral pazopanib hydrochloride once daily for up to 16 weeks in the absence of disease progression or unacceptable toxicity.
  therapeutic conventional surgery: Patients undergo either partial or radical nephrectomy at least 7 days after completion of pazopanib hydrochloride.
Period: Overall Study
Arm/Group | Treatment Group
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 25
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [37 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Could Undergo Partial Nephrectomy After Pazopanib Therapy
Description: The primary end point was the percentage of patients who could undergo partial nephrectomy after pazopanib therapy. A reduction in tumor size, with pazopanib treatment, may permit the use of a partial nephrectomy, as opposed to a radical nephrectomy. This would help preserve additional vascularized parenchyma.
Time Frame: Partial nephrectomy performed after 8 to 16-weeks of pazopanib prescription. The median interval from treatment start to surgery was 10.6 weeks.
Measure: Count of Participants; unit: Participants
Groups:
- Arm I: Patients receive oral pazopanib hydrochloride once daily for up to 16 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo either partial or radical nephrectomy at least 7 days after completion of pazopanib hydrochloride.
  pazopanib hydrochloride: Oral pazopanib hydrochloride once daily for up to 16 weeks in the absence of disease progression or unacceptable toxicity.
  therapeutic conventional surgery: Patients undergo either partial or radical nephrectomy at least 7 days after completion of pazopanib hydrochloride.
Arm/Group | Arm I
Number analyzed (Participants) | 25
Participants | 6

2. Secondary Outcome: Residual Vascularized Parenchyma After Pazopanib Therapy and Subsequent Surgery Relative to Pre-therapy Assessment.
Description: Measurement of total parenchymal tissue that could be saved with pazopanib therapy and subsequent surgery, which was performed via a volumetric analysis of CT images.
Time Frame: After 8 to 16-weeks of pazopanib therapy and 7 day washout prior to surgery.
Measure: Mean (Inter-Quartile Range); unit: cm^3
Arm/Group | Treatment Group
Number analyzed (Participants) | 25
cm^3 | 173 [127 to 238]

3. Secondary Outcome: Change in Tumor Diameter
Description: Median (cm) tumor size reduction after pazopanib treatment, relative to baseline (i.e., before treatment).
Time Frame: At the conclusion of 8 to 16-week treatment with pazopanib therapy.
Measure: Median (Inter-Quartile Range); unit: cm
Groups:
- Treatment Group: Patients receive oral pazopanib hydrochloride once daily for up to 18 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo either partial or radical nephrectomy at least 7 days after completion of pazopanib hydrochloride.
  pazopanib hydrochloride: Oral pazopanib hydrochloride once daily for up to 18 weeks in the absence of disease progression or unacceptable toxicity.
  therapeutic conventional surgery: Patients undergo either partial or radical nephrectomy at least 7 days after completion of pazopanib hydrochloride.
Arm/Group | Treatment Group
Number analyzed (Participants) | 25
cm | 5.5 [1.8 to 8.3]

4. Secondary Outcome: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for Target Lesions: Complete Response, Partial Response, Overall Response (OR)=CR+PR
Description: Efficacy of pazopanib was evaluated via the Response Evaluation Criteria in Solid Tumors, version 1.1. Assessed by MRI. Definitions of response include Complete Response (CR), Disappearance of target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR)=CR+PR
Time Frame: At the end of 8 to 16-weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 25
Participants | 10

5. Secondary Outcome: Surgical Morbidity
Description: Conversion of tumor post therapy so that there is < 10% risk that a partial nephrectomy would be associated with a high risk of significant postoperative morbidity (e.g. conversion of tumor post therapy to ≥ 3 mm away from renal hilum (main renal artery, renal vein, or primary branches)
Time Frame: post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 25
Participants | 16

6. Secondary Outcome: Reduction in Tumor Volume After Treatment
Description: Median (cm^3) tumor size reduction after pazopanib treatment, relative to baseline (i.e., before treatment).
Time Frame: After 8 to 16-weeks of pazopanib treatment
Measure: Mean (Inter-Quartile Range); unit: cm^3
Arm/Group | Treatment Group
Number analyzed (Participants) | 25
cm^3 | 92 [50 to 118]

ADVERSE EVENTS:
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 25/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=25)
Hypertension (Vascular disorders) | 9 — CTCAE grade 3
Elevated Liver Enzymes (Hepatobiliary disorders) | 5 — CTCAE grade 3
Fatigue (General disorders) | 2 — CTCAE grade 3
Thrombocytepenia (Blood and lymphatic system disorders) | 1 — CTCAE grade 3
Fatigue (General disorders) | 19 — CTCAE 1/2
Liver enzymes (Hepatobiliary disorders) | 12 — CTCAE 1/2
Hypertension (Vascular disorders) | 4 — CTCAE 1/2
Diarrhea (Gastrointestinal disorders) | 13 — CTCAE 1/2
Thrombocytopenia (Blood and lymphatic system disorders) | 12 — CTCAE 1/2
Taste Change (General disorders) | 12 — CTCAE 1/2
Nausea/vomiting (Gastrointestinal disorders) | 12 — CTCAE 1/2
Mucositis (Gastrointestinal disorders) | 11 — CTCAE 1/2
Hair Depigmentation (General disorders) | 11 — CTCAE 1/2
Anorexia (Psychiatric disorders) | 11 — CTCAE 1/2
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 9 — CTCAE 1/2
Increased Creatinine (Renal and urinary disorders) | 6 — CTCAE 1/2
Weight Loss (Metabolism and nutrition disorders) | 6 — CTCAE 1/2
Increased Bilirubin (Hepatobiliary disorders) | 5 — CTCAE 1/2

LIMITATIONS AND CAVEATS:
Requires further prospective study. Moreover, in this study, assessment of if partial nephrectomy is feasible prior to surgery was based on subjective measures. Outcome of subjects if they did not receive neoadjuvant therapy is unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No